CLINICAL TRIAL: NCT05468372
Title: A Randomized Controlled Trial of Amphotericin B Versus Posaconazole for Treating Pulmonary Mucormycosis
Brief Title: Amphotericin Versus Posaconazole for Pulmonary Mucormycosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEC-INT/2022/DM-262
Record Dates: First submitted 2022-07-16; First posted 2022-07-21 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Mucormycosis; Pulmonary (Etiology)
Keywords: fungal pneumonia,; zygomycosis; invasive mold disease; Mucorales; Posaconazole
MeSH Terms: conditions — Mucormycosis; Zygomycosis | interventions — posaconazole; liposomal amphotericin B

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amphotericin B arm (standard of care) (Active Comparator): Intravenous liposomal amphotericin B [5 mg/kg per day] for at least 4 weeks followed by maintenance therapy. Maintenance therapy (after four weeks of treatment initiation) will be continued for at least 12 weeks or longer as decided by the treating physician. The maintenance therapy will be posaconazole. However, if therapeutic drug monitoring is not possible or the participants opt to use isavuconazole or amphotericin, the same will be permitted and noted
  Interventions: Drug: Liposomal Amphotericin B
- Posaconazole arm (Experimental): Combination of liposomal amphotericin B (5 mg/kg per day) and posaconazole for first 7 days followed by oral posaconazole only (for induction as well as maintenance therapy). The first four weeks of therapy will be called induction therapy
  Interventions: Drug: Posaconazole 600 mg followed by posaconazole 300 mg once daily; Drug: Liposomal Amphotericin B

INTERVENTIONS:
Drug: Posaconazole 600 mg followed by posaconazole 300 mg once daily — Posaconazole will be given as a delayed release tablet, the dose would be 600 mg in two divided doses on day 1, followed by 300 mg once a day from then on. If a subject vomits within 15 minutes of posaconazole tablet administration, the dosing should be repeated as soon as possible, following appropriate antiemetic treatment. The drug will be administered after a meal.
  Other Names: In the experimental arm, the first seven days of posaconazole will be overlapped with liposomal amphotericin B 5 mg/kg body weight intravenous infusion (similar to the active comparator arm)
  Arms: Posaconazole arm
Drug: Liposomal Amphotericin B — All study subjects will be administered intravenous liposomal amphotericin B [5 mg/kg/day infusion in 5% dextrose solution] over at least 2 hours, as per recommendations. Amphotericin B will be administered for the first seven days in the experimental arm, whereas it will be administered atleast for four weeks in the active comparator arm. Premedication or intravenous hydration will not be routinely administered. For patients experiencing chills, fever, hypotension, nausea, or other non-anaphylactic immediate infusion-related reactions, premedication (acetaminophen, diphenhyramine or hydrocortisone) will be administered 30 to 60 minutes prior to the next dose of amphotericin infusion.
  The dose of intravenous amphotericin B will be modified further if required, based on the tolerability, and response to treatment.
  Other Names: LAMB

SUMMARY:
Pulmonary mucormycosis is a serious illness with high morbidity and mortality (approximately 57%). Surgery and antifungal therapy are central in the management of mucormycosis. Unlike rhino-orbital mucormycosis, surgery is not feasible in several patients with pulmonary mucormycosis. Hence, treatment is primarily with antifungal therapy. Amphotericin B is the standard of care in the medical management of mucormycosis. However, amphotericin B is expensive, has significant adverse events, and is available only in parenteral formulation. Posaconazole is effective against Mucorales, and is currently approved for salvage therapy of mucormycosis. Recent evidence suggest that in several patients, posaconazole may be effective as a monotherapy upfront. In the current study posaconazole versus amphotericin B will be evaluated for the management of pulmonary mucormycosis in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Subjects with proven or probable pulmonary mucormycosis. Participants with a suspicion of pulmonary mucormycosis (as defined previously) based on compatible clinical presentation and compatible imaging will be screened for inclusion in the study.

Exclusion Criteria:

* Failure to provide informed consent
* Contraindications or hypersensitivity to amphotericin B, posaconazole or their components
* Already received >4 days of antifungals prior to randomization into the study
* Pregnant women
* High chances of mortality within 48 hours of enrolment into the study

Subjects with possible pulmonary mucormycosis will also be excluded, if their diagnosis is not confirmed within four working days of enrollment

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants achieving a successful outcome (complete response or partial response) at the completion of six weeks. The response assessment will be a composite of clinical and radiological as adjudged by a multidisciplinary team | six weeks after randomization
  Overall response based on clinical assessment at six weeks after randomization as described recently in a Delphi consensus statement and previous studies on invasive mold infection of the lung. (PMID: 35390293) Based on clinical and radiological response (assessed on CT scan using the two-dimensional measurement of the largest target lesion [WHO criteria, like in lung cancer response assessment]). The overall response will be classified as complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) or death. CR or PR will be labeled success, while SD, PD or death will be labeled as failure

SECONDARY OUTCOMES:
The proportion of participants achieving a successful outcome (complete response or partial response) at the completion of twelve weeks. The response assessment will be a composite of clinical and radiological as adjudged by a multidisciplinary team | telve weeks after randomization
  Overall response based on clinical assessment at twelve weeks after randomization as described recently in a Delphi consensus statement and previous studies on invasive mold infection of the lung. (PMID: 35390293) Based on clinical and radiological response (assessed on CT scan using the two-dimensional measurement of the largest target lesion [WHO criteria, like in lung cancer response assessment]). The overall response will be classified as complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) or death. CR or PR will be labeled success, while SD, PD or death will be labeled as failure
90-day mortality | 90 days after randomization
  Survival at 90 days will be assessed either by in-person or telephonic follow-up
Adverse events related to therapy and the number of participants needing either discontinuation or modification of drug therapy due to adverse events | First four weeks of randomization
  Adverse events to liposomal amphotericin B and posaconazole including deranged liver and renal functions will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided